CLINICAL TRIAL: NCT06883357
Title: The Effects of Home-based Graded Repetitive Arm Supplementary Program Group on Stroke: the Randomized Controlled Trial.
Brief Title: The Effects of Home-based Graded Repetitive Arm Supplementary Program Group on Stroke.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202407010RINB
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRASP group (Experimental)
  Interventions: Behavioral: Graded repetitive arm supplementary program (GRASP)
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Graded repetitive arm supplementary program (GRASP) — Graded repetitive arm supplementary program (GRASP) is a self administrated, home-based rehabilitation program. home-based GRASP program could facilitate the motor function and motor recovery and prevent learned nonuse of affected upper limb of stroke patients. Participants in experimental group will receive Home GRASP program which will be executed 1hour at home per day. In addition, Participants will be requested to return hospital for follow-up and adjusting the training program in group discussion 3 times per week, lasting 4-6 weeks, and totally 12-18 sessions.
  Arms: GRASP group

SUMMARY:
Graded repetitive arm supplementary program (GRASP) is a self administrated, home-based rehabilitation program and has been incorporated in Canadian Stroke Best Practice Recommendations. Past studies indicated that the home-based GRASP program could facilitate the motor function and motor recovery and prevent learned nonuse of affected upper limb of stroke patients. There is lacking of research and application of the home-based GRASP program in Taiwan. Therefore, this study aims to explore the effects of the home-based GRASP program, which is mainly executed in the form of group intervention, on the affected upper limb of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age is above 20 years old.
2. Onset of first stroke complicated with hemiplegia or hemiparesis.
3. The affected upper limb remains partially voluntary movements including lifting to chest level and holding for five seconds; slight flexion and extension of wrist and hand.
4. Understanding and complying with two-steps commands.
5. Understanding the content of trial and willing to sign informed consent.

Exclusion Criteria:

1. Complicating with other neurological disease.
2. Having Orthopedic diseases affecting the movements of upper limbs.
3. Having symptoms of pain to affect the movements of upper limbs.
4. Unstable vital sign or medical condition.
5. Participating another rehabilitative or drug research meanwhile.
6. Receiving botulinum toxin injection within three months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for upper extremity (FMA-UE) | From enrollment to the end of treatment at 6 weeks
  The Fugl-Meyer Assessment for upper extremity (FMA-UE) includes 33 items for the motor recovery of upper limb. Each item is a 3 point ordinal scale. The total score ranges from 0 to 66, higher score means better motor recovery.
Jamar Hydraulic Hand Dynamometer (Jamar Dynamometer) | From enrollment to the end of treatment at 6 weeks
  The Jamar Hydraulic Hand Dynamometer (Jamar Dynamometer) is a tool used for assessing the strength of grip, lateral pinch, and palmar pinch. The muscle strength is recorded in kilograms or pounds.
Action Research Arm Test (ARAT) | From enrollment to the end of treatment at 6 weeks
  The Action Research Arm Test (ARAT) is developed for measuring the motor function of affected upper limb after stroke. ARAT includes subscales of grasp, grip, pinch, and gross movement. The total score ranges from 0 to 57, higher score means better motor function.

SECONDARY OUTCOMES:
Chedoke Arm and Hand Activity Inventory (CAHAI) | From enrollment to the end of treatment at 6 weeks
  The Chedoke Arm and Hand Activity Inventory (CAHAI) is developed for measuring the level of function and involvement of the affected upper limb in bimanual tasks. It contains 13 tasks and the total score is ranged from 13 to 91. The higher score means better motor function and involvement.
Rating of Everyday Arm-use in the Community and Home Scale (REACH-Scale) | From enrollment to the end of treatment at 6 weeks
  The Rating of Everyday Arm-use in the Community and Home Scale (REACH-Scale) is a self-evaluation scale designed for stroke patients to measure the involvement of the affected upper extremity in everyday life. The score ranged from 0 to 5 and higher score indicate the more utilization of affected upper extremity.
Stroke Impact Scale Version 3.0 (SIS 3.0) | From enrollment to the end of treatment at 6 weeks
  The Stroke Impact Scale Version 3.0 (SIS 3.0) is a self-evaluated assessment for measuring the quality of life of patients with stroke. In our study, the strength domain(total score:4-20) and hand function domain(total score:5-25), and the an extra question on stroke recovery(total score:0-100)was used. The higher score means better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yi Lin, Study Director — Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No